CLINICAL TRIAL: NCT01891526
Title: The Pharmacokinetics of a Single Dose of 9-cis-retinoic Acid (Alitretinoin, Toctino®) in Patients With Moderate to Severe Hepatic Insufficiency
Brief Title: Single Dose of 9-cis-retinoic Acid in Hepatic Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Frederik Grønlund MD DMSci, MD, University Hospital, Gentofte, Copenhagen
Other Study IDs: 2010-338; Allitretinoin
Record Dates: First submitted 2013-06-21; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: Hepatic Insufficiency
Keywords: Metabolisation of 9-cis-retinoic acid; hepatic patients; investigation of urine and blood samples
MeSH Terms: conditions — Hepatic Insufficiency | interventions — Alitretinoin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hepatic patients: patients with hepatic insufficiency
  Interventions: Drug: 9-cis-retinoic acid
- Healthy Controls: Healthy adults
  Interventions: Drug: 9-cis-retinoic acid

INTERVENTIONS:
Drug: 9-cis-retinoic acid — Single dose of 9-cis-retinoic acid (Capsule 30 mg) as oral exposure

SUMMARY:
To test whether patients with hepatic insufficiency can tolerate one oral dose of 9-cis-retinoic acid and to test whether the metabolism of retinoic acid is altered.

ELIGIBILITY:
Inclusion Criteria:

1. Have biopsy verified hepatic insufficiency
2. Medically stable.
3. Ultra sonic examination of lever within the past 3 months
4. No pregnancy documented in women. use of anticonception during study and 1 month after

Exclusion criteria:

1. Odd blood counts and samples not related to hepatic disease
2. encephalopathy (> grad II)
3. concomitant treatment with pharmaca that is metabolized by CYP3A4 in the liver.
4. Cardiac disease
5. Kidney disease
6. Epilepsia
7. Stroke
8. Esophagal bleeding
9. Severe ascites
10. HIV-positivity
11. Psychiatric disorder
12. Cancer
13. pregnancy or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 patients with hepatic disease and 10 controls
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
A comparison of the metabolisation of retinoic acid in patients with hepatic insufficiency and controls | 24 hours
  Analysis on samples

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Gentofte Municipality, Denmark